CLINICAL TRIAL: NCT04917718
Title: Assessment of Renal Tubular Injury and Transplant Outcomes in Cardiac Recipients Converting From Immediate Release Tacrolimus to Extended Release Tacrolimus.
Brief Title: Renal Tubular Injury and Transplant Outcomes in Cardiac Recipients Converting From IR Tacrolimus to XR Tacrolimus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sanjeev Akkina, MD, Associate Professor of Medicine, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 212781
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Diseases; Heart Transplant
Keywords: Immediate Release Tacrolimus; Extended Release Tacrolimus; IR Tacrolimus; XR Tacrolimus; Renal Tubular Injury; Heart Transplant Recipient; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Extended Release Tacrolimus (Experimental): All participants who consent to the study will be in this group.
  Interventions: Drug: Conversion from IR Tacrolimus to XR Tacrolimus

INTERVENTIONS:
Drug: Conversion from IR Tacrolimus to XR Tacrolimus — All participants will be consented to the study on IR Tacrolimus. After their baseline visit, they will be converted to XR Tacrolimus

SUMMARY:
Immediate release (IR) tacrolimus peaks in the first two hours after administration. These peak levels are influenced by CYP3A5 expression with expressors requiring higher total daily doses with higher peak levels compared to non-expressors. Tacrolimus XR (Envarsus) is a once daily formulation with delayed absorption and lower peak levels while maintaining similar trough levels as seen with IR tacrolimus. A randomized trial of conversion from IR tacrolimus to tacrolimus XR in kidney transplant recipients have shown similar efficacy and adverse events between the two groups but no improvement in estimated GFR. However, urinary biomarkers of acute kidney injury associated with changes in tacrolimus dosing may be more sensitive then serum creatinine. The objective of this study is to assess renal tubular injury in heart transplant recipients who are converted from immediate release to tacrolimus XR. The hypothesis is that the delayed absorption and lower peak levels of tacrolimus XR will lead to less tubular injury and improved renal function without increased risk to the heart allograft.

DETAILED DESCRIPTION:
The primary outcome is change in urinary NGAL expression with conversion from IR tacrolimus to tacrolimus XR. In aim 1, changes in urinary biomarkers of tubular injury at 4 weeks after conversion to tacrolimus XR with stable trough levels will be assessed. These changes will be assessed by CYP3A5 expressor category that will be determined by genotyping of a single gene for variants. The changes in GFR using the creatinine-cystatin C CKD-EPI equation will be assessed. In aim 2, the rate of rejection as defined as treated rejection within the last 30 days for any grade > 1R or AMR or acute graft dysfunction (LV ejection fraction drop > 10%) will be looked. The cardiac allograft vasculopathy based on coronary angiography +/- IVUS and right heart catheterization hemodynamics at baseline and 1 year post conversion will also be evaluated. In addition to changes in cardiac function, the changes in blood pressure, serum glucose, and cholesterol in the first year after conversion will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Stable, heart-only transplant recipient within 10 years of transplantation
* 18 -80 years old
* Currently taking IR Tacrolimus
* Baseline eGFR> 30mL/min/1.73m2

Exclusion Criteria:

* Multiple organ transplant recipients
* Less than 18 years old
* Greater than 80 years old
* Heart-only transplants recipients with active malignancy, rejection, or greater than 10 years from transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary neutrophil gelatinase-associated lipocalin (NGAL) | 4 weeks
  Change in Urinary NGAL level (ng/mL)

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate (eGFR) | 4 weeks
  Change in eGRF level by the Creatinine-Cystatin C CKD-EPI equation (mL/min/1.73m2)
Microalbuminuria | 4 weeks
  Change in Urine albumin-creatinine ratio
CYP3A5 expressor category | Baseline
  CYP3A5 genotyping to determine expressor category
Heart transplant rejection | 1 year
  The rate of rejection as defined as treated rejection within the last 30 days for any grade>1R, AMR, or acute graft dysfunction (LVEF drop greater than 10%)
Cardiac allograft vasculopathy | 1 year
  The rate of cardiac allograft vasculopathy based on coronary angiography with or without IVUS and right heart catheterization hemodynamics
Blood pressure | 1 year
  Change in blood pressure (mmHg)
Serum glucose | 1 year
  Change in serum glucose levels (mg/dL)
LDL Cholesterol | 1 year
  Change in LDL cholesterol level (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Akkina, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ojo AO, Held PJ, Port FK, Wolfe RA, Leichtman AB, Young EW, Arndorfer J, Christensen L, Merion RM. Chronic renal failure after transplantation of a nonrenal organ. N Engl J Med. 2003 Sep 4;349(10):931-40. doi: 10.1056/NEJMoa021744. PMID 12954741
- [Background] Naesens M, Kuypers DR, Sarwal M. Calcineurin inhibitor nephrotoxicity. Clin J Am Soc Nephrol. 2009 Feb;4(2):481-508. doi: 10.2215/CJN.04800908. PMID 19218475
- [Background] Camara NO, Matos AC, Rodrigues DA, Pereira AB, Pacheco-Silva A. Early detection of heart transplant patients with increased risk of ciclosporin nephrotoxicity. Lancet. 2001 Mar 17;357(9259):856-7. doi: 10.1016/S0140-6736(00)04207-0. PMID 11265958
- [Background] Myers BD, Ross J, Newton L, Luetscher J, Perlroth M. Cyclosporine-associated chronic nephropathy. N Engl J Med. 1984 Sep 13;311(11):699-705. doi: 10.1056/NEJM198409133111103. PMID 6382005
- [Background] Cosio FG, Amer H, Grande JP, Larson TS, Stegall MD, Griffin MD. Comparison of low versus high tacrolimus levels in kidney transplantation: assessment of efficacy by protocol biopsies. Transplantation. 2007 Feb 27;83(4):411-6. doi: 10.1097/01.tp.0000251807.72246.7d. PMID 17318073
- [Background] Trofe-Clark J, Brennan DC, West-Thielke P, Milone MC, Lim MA, Neubauer R, Nigro V, Bloom RD. Results of ASERTAA, a Randomized Prospective Crossover Pharmacogenetic Study of Immediate-Release Versus Extended-Release Tacrolimus in African American Kidney Transplant Recipients. Am J Kidney Dis. 2018 Mar;71(3):315-326. doi: 10.1053/j.ajkd.2017.07.018. Epub 2017 Nov 20. PMID 29162334
- [Background] Bunnapradist S, Ciechanowski K, West-Thielke P, Mulgaonkar S, Rostaing L, Vasudev B, Budde K; MELT investigators. Conversion from twice-daily tacrolimus to once-daily extended release tacrolimus (LCPT): the phase III randomized MELT trial. Am J Transplant. 2013 Mar;13(3):760-9. doi: 10.1111/ajt.12035. Epub 2012 Dec 21. PMID 23279614
- [Background] Chancharoenthana W, Leelahavanichkul A, Wattanatorn S, Avihingsanon Y, Praditpornsilpa K, Eiam-Ong S, Townamchai N. Alteration of urinary neutrophil gelatinase-associated lipocalin as a predictor of tacrolimus-induced chronic renal allograft fibrosis in tacrolimus dose adjustments following kidney transplantation. PLoS One. 2018 Dec 21;13(12):e0209708. doi: 10.1371/journal.pone.0209708. eCollection 2018. PMID 30576367
- [Background] Vaidya VS, Ozer JS, Dieterle F, Collings FB, Ramirez V, Troth S, Muniappa N, Thudium D, Gerhold D, Holder DJ, Bobadilla NA, Marrer E, Perentes E, Cordier A, Vonderscher J, Maurer G, Goering PL, Sistare FD, Bonventre JV. Kidney injury molecule-1 outperforms traditional biomarkers of kidney injury in preclinical biomarker qualification studies. Nat Biotechnol. 2010 May;28(5):478-85. doi: 10.1038/nbt.1623. PMID 20458318
- [Background] Tsuchimoto A, Shinke H, Uesugi M, Kikuchi M, Hashimoto E, Sato T, Ogura Y, Hata K, Fujimoto Y, Kaido T, Kishimoto J, Yanagita M, Matsubara K, Uemoto S, Masuda S. Urinary neutrophil gelatinase-associated lipocalin: a useful biomarker for tacrolimus-induced acute kidney injury in liver transplant patients. PLoS One. 2014 Oct 20;9(10):e110527. doi: 10.1371/journal.pone.0110527. eCollection 2014. PMID 25329716